CLINICAL TRIAL: NCT06917859
Title: Prophylactic Methylprednisolone for Renal Protection in Cardiac Surgeries With Cardiopulmonary Bypass: A Randomized Double-Blinded Clinical Study
Brief Title: Prophylactic Methylprednisolone for Renal Protection in Cardiac Surgeries With Cardiopulmonary Bypass
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD47/2025
Record Dates: First submitted 2025-02-14; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: Cardiopulmonary Bypass; AKI - Acute Kidney Injury
Keywords: AKI; CPB
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): (Placebo group / Control group) will receive normal saline as a placebo after the induction of anesthesia and before initiating CPB.
- Methylprednisolone group (Active Comparator): (Methylprednisolone group ) receive a single intra-venous dose of methylprednisolone (2 mg/kg) after the induction of anesthesia, and before the initiation of CPB.
  Interventions: Drug: Methylprednisolone group

INTERVENTIONS:
Drug: Methylprednisolone group — In this study patients will be given a single intra-venous dose of methylprednisolone (2 mg/kg) after the induction of anesthesia, and before the initiation of CPB.
  Arms: Methylprednisolone group

SUMMARY:
The aim of the planned study is to assess the prophylactic effect of intraoperative administration of a single dose of methylprednisolone 2 (mg/kg) in decreasing the incidence of postoperative acute kidney injury after cardiac surgeries with cardiopulmonary bypass.

DETAILED DESCRIPTION:
Patients undergoing any type of elective cardiac surgical procedure requiring CPB will be randomly assigned into one of the following groups

1. Placebo group / Control group will receives normal saline as a placebo after the induction of anesthesia and before initiating CPB.
2. Methylprednisolone group / Interventional group receives a single intra-venous dose of methylprednisolone (2 mg/kg) after the induction of anesthesia, and before the initiation of CPB.

Measurements:

Primary outcome:

Incidence of occurrence of postoperative acute kidney injury for 7 days according to the RIFLE criteria.

Secondary outcome:

1. Incidence of postoperatively hyperglycemia (blood glucose level of ≥ 140 mg/dl) for 7 days,
2. Duration of ICU stay,
3. Length of hospital stay (LOS),
4. Incidence of wound infection,
5. Incidence of peptic ulcer,
6. Incidence of sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Sex: Both sexes.
3. Patients with American Society of Anesthesiologists (ASA) score III-IV.
4. Patients scheduled for any kind of elective cardiac surgical procedure requiring cardiopulmonary bypass (e.g., coronary artery bypass grafting (CABG), valve repair/replacement, or combined procedures (

Exclusion Criteria:

1. Declining to give written informed consent.
2. History of allergy to the medications used in the study.
3. Diabetic patients with HbA1C >6.5
4. Moderate to severe hepatic diseases (Child B-C)
5. Hepatic dysfunction: INR > 1.5, serum albumin < 2.9 g%.
6. Renal dysfunction (serum Creatinine level >1.3 mg/dl, or GFR < 80 ml/min./1.73/m2
7. Patients with a recent history of AKI.
8. Patients undergoing urgent cardiac surgery.
9. Patients undergoing cardiac surgeries with deep hypothermic total circulatory arrest.
10. Planned off-pump procedure.
11. Any cardiac surgery exceeds 45 minutes on Aortic cross clamp.
12. Patients requiring high doses of inotropes and/or vasopressors intraoperative or postoperative (high-dose dopamine is defined as peak doses of >15 μg/kg/min, high-dose norepinephrine is defined as peak dose >0.1 μg/kg/min, high-dose epinephrine is defined as peak dose >0.1 μg/kg/min)
13. Delayed extubation for more than 6 hours postoperative.
14. Patients developed postoperative complications as (septic shock and bleeding)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of occurrence of postoperative acute kidney injury | 7 days post-operative
  Incidence of occurrence of postoperative acute kidney injury for 7 days according to the RIFLE criteria.

SECONDARY OUTCOMES:
Incidence of postoperatively hyperglycemia | 7 days post-operative
  1. Incidence of postoperatively hyperglycemia (blood glucose level of ≥ 140 mg/dl).
Duration of ICU stay, | 7 days post-operative
  Duration of ICU stay,
Length of hospital stay | 14 Day post-operative
  Length of hospital stay
Incidence of wound infection | 7 days post-operative
  Incidence of wound infection
Incidence of peptic ulcer | 7 days post-operative
  Monitoring attacks of hematemesis or melena
Incidence of sepsis | 7 days post-operative
  Incidence of sepsis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt